CLINICAL TRIAL: NCT04644380
Title: Assessment of the INVOcell Culture Device When Used for up to Five-Day Incubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INVO Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-018
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): During an IVF/IVC cycle, participants will retain the INVOcell Culture Device with the Retention Device in the vaginal cavity for 5 days vaginal incubation
  Interventions: Device: INVOcell

INTERVENTIONS:
Device: INVOcell — Female participants undergoing in vitro fertilization (IVF) and or/or Intracytoplasmic Sperm Injection (ICSI) for assisted reproductive will be asked to participate
  Other Names: Intravaginal Culture; IVC; Vaginal incubation

SUMMARY:
The INVOcell Culture Device received de novo request for 3-day intravaginal incubation. The device is held in place with the intravaginal cavity by a Retention Device. The clinical study will assess the ability of a modified Retention Device to hold INVOcell in place during 5-day vaginal incubation as well as comfort and vaginal irritation as secondary endpoints.

DETAILED DESCRIPTION:
This is a single center, open label non-comparative prospective trial to evaluate the retention of the INVOcell IVC with the Retention Device over the vaginal incubation period of up to 5 days.

The purpose of this study is to assess the retention of the INVOcell IVC device with the Retention Device over the vaginal incubation period of up to 5 days.

Primary Endpoint

• Retention of the INVOcell IVC device with the Retention Device over the vaginal incubation period of up to 5 days.

Secondary Endpoint

* Comfort of the INVOcell IVC and Retention Device
* Vaginal tissue reactions during the vaginal incubation
* Optical clarity and the ability to visualize the embryos after the incubation

ELIGIBILITY:
Inclusion Criteria:

* Have been informed about the study and have given their written consent.
* Patients 18 years to 42 years
* Women who are scheduled for an oocyte retrieval in anticipation of INVOcell IVF.

Exclusion Criteria:

* Inability to read and speak English fluently
* Identified vaginal infection
* Recent pelvic surgery based on clinical history and physical examination.
* History of toxic shock syndrome
* Inability to tolerate the placement or wearing of the INVOcell IVC or INVOcell Retention Device.
* Inability to tolerate a speculum examination
* Unwilling or unable to wear the INVO Retention (diaphragm) during the incubation.
* Unable or unwilling to sign informed consent or abide by study follow up assessment requirements.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Device Retention | 5 days
  The primary endpoint is INVOcell IVC retention with the Retention Device. The following will be assessed:
  Whether the INVOcell IVC stays in place (is retained within the vaginal cavity) while being used with the Retention Device during 5 days of continuous vaginal incubation.

SECONDARY OUTCOMES:
Comfort | 5 days
  Comfort of the INVOcell IVC while worn with the Retention Device evaluated on a 10-oint Likert scale.
Vaginal tissue reactions | 5 days
  Vaginal tissue reactions during the vaginal incubation based on post removal and assessed by vaginal speculum examination performed to examine the vaginal walls speculum examination post removal vaginal examination.
Optical clarity | 5 days
  Optical clarity and the ability to visualize the embryos after the incubation of the INVOcell device.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hammond, DNP, CRNP, Principal Investigator — American Institute of Reproductive Medicine/IVD Alabama (AIRM)
Locations (1):
- American Institute of Reproductive Medicine/IVF Alabama (AIRM), Homewood, Alabama, United States

IPD SHARING:
Plan to Share IPD: No